CLINICAL TRIAL: NCT07158671
Title: The Effectiveness of the mHealth Survivorship Program on Enhancing Health-related Quality of Life Among Colorectal Cancer Survivors: Randomised Controlled Trial
Brief Title: The Effectiveness of the mHealth Survivorship Program on Enhancing Health-related Quality of Life Among Colorectal Cancer Survivors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Nethersole School of Nursing (Other)
Responsible Party: Principal Investigator, Do Pham Nhat Vi, PhD Candidate, The Nethersole School of Nursing
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025.327
Record Dates: First submitted 2025-08-19; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer (Diagnosis)
Keywords: mHealth; Survivorship; Colorectal cancer; Survivors; health-related quality of life
MeSH Terms: conditions — Colorectal Neoplasms; Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Participants in the control group will receive the usual care
- mHealth survivorship program (Active Comparator): Participants in the intervention group will:
  Use the survivorship programme through mHealth every day for 3 months; Be called by the healthcare provider every 2 weeks for consultation
  Interventions: Other: Intervention Group

INTERVENTIONS:
Other: Intervention Group — Participants in the intervention group will:
  Use the survivorship programme through mHealth every day for 3 months; Be called by the healthcare provider every 2 weeks for consultation
  Arms: mHealth survivorship program

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of the mHealth survivorship program in enhancing health-related quality of life among colorectal cancer survivors. It is hypothesized that participants receiving the mHealth-based survivorship program will report significantly higher levels of health-related quality of life and a lower level of distress, depression, anxiety, fatigue, and bowel dysfunction compared to those in the control group.

Participants in the intervention group will:

Use the survivorship programme through mHealth every day for 3 months Be called by the healthcare provider every 2 weeks for consultation

Participants in the control group will receive the usual care

DETAILED DESCRIPTION:
Cancer is the second leading cause of global mortality, with colorectal cancer (CRC) ranking third in deaths and diagnoses for both genders. There are more and more survivors who have completed treatment, improving survival rates and emphasizing the need for ongoing support. CRC survivors face challenges due to a lack of healthcare support, which can reduce their quality of life (QoL). The Institute of Medicine (IOM) recommends specialized survivorship programmes for CRC survivors. The American Cancer Society (ACS) has also issued comprehensive guidelines for CRC survivorship care. Evidence suggests that integrating a mobile application can improve resource coordination for survivors in remote areas, enhancing QoL. Thus, developing mHealth-based survivorship programs aligned with ACS guidelines is crucial for improving health-related QoL in this population.

Briefly, as a result of a systematic review and meta-analysis, we identified two key features of the available survivorship programmes and their efficacy in enhancing health-related QoL. First, many programmes have methodological weaknesses, with few studies adequately reporting allocation concealment or non-blinding. Only 7 out of 22 studies were grounded in different theoretical frameworks, and none were conducted in developing countries. Second, each programme was often treated in isolation, and the contents followed the ACS guidelines. They emphasise health promotion and managing late side effects over surveillance for second cancers and care coordination. Key components include: 1) CRC education on symptom management, nutrition, and exercise; 2) expert health coaching with survivorship care plans, delivered over 12 weeks, averaging 30-45 minutes, 6 to 12 sessions weekly; delivered mobile health, led by nurses. From these gaps, rigorous studies are warranted to integrate these contents to lay the foundation for future comprehensive interventions via mobile health, which can address multiple domains to improve the health-related QoL for this population.

This study will adopt a randomised controlled trial (RCT) design. A total of 210 participants will be recruited, including 50 participants for pilot RCT and 160 participants for the main RCT. Participants in the intervention group will receive the mHealth survivorship programme, and participants in the control group will receive usual care. Outcomes will be measured at four timepoints: recruitment (T0), immediately post-intervention (T1), 1-month follow-up (T2). For data analysis, ITT analyses will be conducted. All the statistical analyses will be performed via R, and the significance level of 0.05 will be set.

ELIGIBILITY:
Inclusion Criteria:

* be 18 or older (1);
* Vietnamese-speaking CRC patients who have completed active treatment and are preparing for discharge (2);
* provide consent and complete questionnaires independently (3);
* no metastatic and second cancers (4);
* using the Android smartphone (5).

Exclusion Criteria:

* mental health diseases;
* receiving anxiety or depression treatment or cognitive/learning problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
The Functional Assessment of Cancer Therapy-General (FACT-G) | Participants will be assessed at three-time points: baseline (Day 1), post-intervention (12 weeks), and 1-month follow-up (after post intervention))
  Assesses health-related QoL, including physical function (consisting of 7 items), social and family relationships (7 items), emotional state (6 items), and functional abilities (7 items). Scores range from 0 to 100, with higher scores indicating better QoL. Cronbach's alpha of 0.89 for the scale, received the approval to use the FACT-G from the FACIT organisation

SECONDARY OUTCOMES:
The distress thermometer screening tool (DT) | Participants will be assessed at three-time points: baseline (Day 1), post-intervention (12 weeks), and 1-month follow-up (after post intervention))
  A self-report tool measuring distress on a scale from 0 (no distress) to 10 (extreme distress), focusing on a cutoff score of 4
The Depression Anxiety Stress Scales (DASS-21) | Participants will be assessed at three-time points: baseline (Day 1), post-intervention (12 weeks), and 1-month follow-up (after post intervention))
  Consists of 21 items, with seven items for anxiety (DASS21-A), seven items for depression (DASS21-D) and seven items for stress (DASS21-S). It was validated for use in the Vietnamese population with good internal consistency (Cronbach's alpha: depression subscale-0.72; anxiety subscale-0.77; stress subscale-0.70, and overall scale-0.88).
The Functional Assessment of Cancer Therapy-Fatigue subscale (FACT-F) | Participants will be assessed at three-time points: baseline (Day 1), post-intervention (12 weeks), and 1-month follow-up (after post intervention))
  with 13 items, likert scales from 0 (not at all) to 4 (ver much), which has been validated for use in the Vietnamese version with Cronbach's alpha coefficient α = 0.93
The Low anterior resection syndrome (LARS) | Participants will be assessed at three-time points: baseline (Day 1), post-intervention (12 weeks), and 1-month follow-up (after post intervention))
  A 5-question questionnaire evaluated bowel functional symptoms. Scores were assigned to responses, determining the LARS score, which categorized results into "no LARS" (0-20), "minor LARS" (21-29), and "major LARS" (30-42). Cronbach's alpha was from 0.874 to 0.934

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-07-04): https://cdn.clinicaltrials.gov/large-docs/71/NCT07158671/Prot_SAP_000.pdf
  • Informed Consent Form (2025-08-15): https://cdn.clinicaltrials.gov/large-docs/71/NCT07158671/ICF_001.pdf